CLINICAL TRIAL: NCT06975761
Title: A COMPARATIVE EVALUATION OF POST-OPERATIVE PAIN AFTER ROOT CANAL THERAPY USING TWO DIFFERENT ENDODONTIC SEALERS IN PATIENTS WITH SYMPTOMATIC IRREVERSIBLE PULPITIS
Brief Title: Postoperative Pain Comparison of Two Root Canal Sealers in Irreversible Pulpitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Armed Forces Institute of Dentistry, Pakistan (Other)
Responsible Party: Principal Investigator, Areeba Maryam, Resident operative dentistry and endodontics, Armed Forces Institute of Dentistry, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pulpdent Versus Ad-seal
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Post Operative Pain After Root Canal Therapy
Keywords: post operative pain; irreversible pulpitis; endodontic sealers
MeSH Terms: conditions — Pain, Postoperative | interventions — epoxy resin-based root canal sealer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Resin based sealer (Active Comparator): Endodontic sealer AD seal and core obturating material single cone F2 gutta parcha(Bio GP points-sure endo, sure dent cooperation)
  Interventions: Drug: Resin Based sealer
- ZnO eugenol based sealer (Active Comparator): Endodontic sealer pulp-dent sealer and core obturating material single cone F2 gutta parcha. (Bio GP points-sure endo, sure dent cooperation)
  Interventions: Drug: ZnO eugenol based sealers

INTERVENTIONS:
Drug: Resin Based sealer — Post-operative pain after Root Canal Therapy by using resin based sealer
  Arms: Resin based sealer
Drug: ZnO eugenol based sealers — Post-operative pain after Root Canal Therapy by using ZnO eugenol based sealer
  Arms: ZnO eugenol based sealer

SUMMARY:
This study, approved by the Institutional Ethics Review Committee, AFID (Annex "A"), will involve 62 eligible patients from the Operative Dentistry Department, Armed Forces Institute of Dentistry. Patients (and their guardians) will receive a detailed explanation in Urdu, and written informed consent will be obtained (Annex "B").

Study Design:

Randomized Controlled Trial: Patients will be randomly divided into two equal groups using a scientific random number table.

Inclusion Screening: Includes medical history, clinical examination, periapical radiographs.

Treatment Protocol:

Root canal therapy under local anesthesia with rubber dam isolation.

Working length determined using DentaPort ZX apex locator, confirmed with radiograph.

Instrumentation: ProTaper Universal hand files up to F2 with 5.25% NaOCl irrigation.

Patency confirmed with #10 K-file between each instrument change.

Final flush with 17% EDTA.

Calcium hydroxide used as intracanal medicament for microbial control.

Temporary restoration using Cavit.

Recall and Evaluation: After 1 week, asymptomatic patients (VAS score 0 and dry canals) will be selected for obturation.

Obturating Materials:

Group 1: AD Seal + F2 single cone gutta-percha (Sure Endo). Group 2: Pulp-dent Sealer + F2 single cone gutta-percha (Sure Endo). Sealers will be mixed per manufacturer's instructions, applied using lentulospiral. The apical extent of the master cone will be confirmed radiographically.

All procedures will be carried out by a single operator. Final restoration will be done using composite, and patients will be referred for full coverage crowns.

Post-Treatment Pain Assessment:Patients will receive a pain diary with a Visual Analogue Scale (VAS) from 0 (no pain) to 10 (severe pain).

Pain will be recorded at 24 hours, 72 hours, and 7 days post-treatment. Analgesic use (type and quantity) will also be noted. Diaries will be collected at the follow-up visit.

DETAILED DESCRIPTION:
Study will be conducted after the approval of Institutional Ethics Review Committee, AFID (ANX "A").

A total of 62 entitled patients reporting to Operative Dentistry Department, Armed Forces Institute of Dentistry will be invited for participation in this study. The procedure will be explained to the patients and their parents in Urdu language and a written informed consent will be taken (ANX "B") Patients will be randomly divided into two equal groups with the help of scientific random number table. They will be screened for inclusion by taking history, performing relevant clinical examination and necessary tests along with peri-apical radiographs. Root canal therapy will be then be initiated under local anaesthesia and rubber dam isolation. Working length will be taken 1mm short of radiographic apex with apex locator (Denta Port ZX) and will be confirmed with radiograph. The root canals will be instrumented with ProTaper Universal hand files (dentsply sirona) under copious irrigation with 5.25% sodium hypochlorite (NaOCl) (vista dental products) up to F2 protaper file(dentsply,sirona) . Patency will be confirmed with a #10 K file (dentsply maillefer) between each instrument change. The root canals will be flushed with of 17% EDTA solution (techno dent edetect gel). To control the microbiological impact on post-operative pain calcium hydroxide will be used as an intra-canal medicament and likewise 5.25% sodium hypochlorite as an irrigant in both groups.

After chemomechanical preparation the canals will be dried using sterile paper points (sure endo) and freshly mixed calcium hydroxide paste will be placed into the prepared canals using a lentulospiral (MAN.inc) which is followed by temparory restoration, cavit (provis). The patients will be recalled after a week and patients who will be asymptomatic exhibiting a VAS Score of 0 and dry canals on evaluation with sterile paper points after removal of the intracanal medicament will be obturated. The teeth will be obturated according to the randomly allocated groups, Group 1: endodontic sealer AD seal and core obturating material single cone F2 gutta parcha(Bio GP points-sure endo, sure dent cooperation).

Group 2: endodontic sealer pulp-dent sealer and core obturating material single cone F2 gutta parcha. (Bio GP points-sure endo, sure dent cooperation).

Manufacturer's instructions will be followed for mixing the respective sealer on a sterile glass slab. The apical extent of the master cone will be confirmed radiographically. The canals will be coated with the sealer using lentulospiral (MAN,Inc.) in a slow speed hand piece followed by the obturation of canals with single cone F2 gutta parcha (Bio GP points-sure endo, sure dent cooperation).

All the clinical procedures will be performed by single operator. After obturation access cavity is restored with composite and the patient will be refered to prosthodontic department for the provision of full coverage crowns.

Post-treatment pain assessment:

After obturation and restoration with composite all the patients will handed over a pain diary form with visual analogue scale (VAS) consisting of a 10 cm line divided into 10 equal parts from 0 indicating no pain to 10 indicating extremely severe pain. This provided a range of score from 0-10. The patients will be asked to record their pain response at 24 hrs, 72 h and 7 days after therapy followed by which the patients will be recalled to give the diary to the investigators on their follow up visit. In case of consumption of analgesics, the type and quantity after treatment will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Permanent mandibular first molar with irreversible pulpitis without swelling and sinus.
2. Patients of male gender between 20-40 years of age.
3. Systemically healthy patients with no other co morbidity classified as ASA-I
4. Patients who agree to attend for re call appointments and provide a written consent

Exclusion Criteria:

- 1. Teeth with calcified canals and previously treated teeth. 2. Mandibular molars with reversible pulpitis. 3. Pregnant and lactating mothers. 4. Patients who are immunocompromised, anxious, mentally ill. 5. Cases of root fracture. 6. Patients who consumed analgesics 12-24 hrs before primary root canal therapy.

7. Patients who are allergic to any of the medications being tested.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-08-07 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Post-Operative pain by using resin based sealer on visual analogue scale | 24 hours
  endodontic sealer AD seal and core obturating material single cone F2 gutta parcha(Bio GP points-sure endo, sure dent cooperation),post-operative pain on visual analogue scale.
Post-Operative pain by using resin based sealer on visual analogue scale | 72 hours
  endodontic sealer AD seal and core obturating material single cone F2 gutta parcha(Bio GP points-sure endo, sure dent cooperation),post operative pain on visual analogue scale
Post-Operative pain by using resin based sealer on visual analogue scale | 7 days
  endodontic sealer AD seal and core obturating material single cone F2 gutta parcha(Bio GP points-sure endo, sure dent cooperation),post operative pain on visual analogue scale
Post-Operative pain by using ZnO engenol based sealer on visual analogue scale | 24 hours
  endodontic sealer pulp-dent sealer and core obturating material single cone F2 gutta parcha. (Bio GP points-sure endo, sure dent cooperation),post-operative pain on visual analogue scale.
Post-Operative pain by using ZnO engenol based sealer on visual analogue scale | 72 hours
  endodontic sealer pulp-dent sealer and core obturating material single cone F2 gutta parcha. (Bio GP points-sure endo, sure dent cooperation),post-operative pain on visual analogue scale
Post-Operative pain by using ZnO engenol based sealer on visual analogue scale | 7 days
  endodontic sealer pulp-dent sealer and core obturating material single cone F2 gutta parcha. (Bio GP points-sure endo, sure dent cooperation),post-operative pain on visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Areeba Maryam, BDS, Principal Investigator — AFID
Locations (1):
- Armed Forces Institute of Dentistry, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided